CLINICAL TRIAL: NCT04391556
Title: Interest of PET-PSMA Imaging Potentiated by Androgen Blockade in Patients With Biological Relapse or Persistent Biological Disease of a Localized Prostatic Adenocarcinoma After Initial Treatment
Brief Title: Interest of PET-PSMA Imaging Potentialised by Androgen Blockade in Localized Prostatic Adenocarcinoma
Acronym: PREFAcE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET19-194 - PREFAcE
Record Dates: First submitted 2020-04-23; First posted 2020-05-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-04

CONDITIONS: Prostate Adenocarcinoma
Keywords: Prostate adenocarcinoma; TEP PSMA; Androgenic blockade
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Firmagon (Experimental): 120 mg Firmagon subcutaneous injection after a TEP-PSMA
  Interventions: Drug: Firmagon

INTERVENTIONS:
Drug: Firmagon — 120 mg subcutaneous Injection of Firmagon after a TEP-PSMA
  Other Names: Injection of Firmagon after a TEP-PSMA

SUMMARY:
Evaluation of the interest of PET-PSMA imaging potentiated by androgen blockade in patients with biological relapse or persistent biological disease of a localized prostatic adenocarcinoma after initial treatment

DETAILED DESCRIPTION:
The identification of lesions responsible for biological recurrence or persistent biological disease in patients with prostatic adenocarcinoma (PA) remains an outstanding problem due to the lack of sensitivity of standard imaging techniques. The efficacy of empirical radiation therapy of the prostate + pelvis zone in only half of patients with increased PSA suggests an underestimation of lesions.

PET-68Ga-PSMA or PET-PSMA technique showed a clear gain in sensitivity for the detection of lesions in this context compared to PET-Choline which was already more sensitive than standard imaging. It is about 50% for a PSA <0.5 ng / ml vs 20% for a PSA <1 ng / ml for TEP-Choline technique. However, the indication of empirical radiotherapy is raised when the PSA exceeds 0.2 ng / ml. It is therefore still necessary to increase the sensitivity of PET-PSMA.

A flare-up-related effect was observed in a small animal experiment and in a patient after androgen blocking treatment, inducing a sharp increase in the intensity of previously visualized lesions and the appearance of 13 new lesions.

It would therefore be possible to increase the expression of PSMA by the lesions at the origin of the biological recurrence of AP and thus to improve their detection by PET-PSMA after potentiation by short-term androgen blocking by an antagonist of LH-RH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Hormone-naive patients, initially treated curatively by prostatectomy for prostate adenocarcinoma and having a first or new biological recurrence (PSA greater than 0.2 ng/ml; confirmed on at least two successive dosages in the last 12 months) OR Hormone-naive patients, initially treated curatively by external radiotherapy or by brachytherapy for prostate adenocarcinoma and having a biological recurrence (PSA Nadir + 2ng/ml ; confirmed on at least two successive dosages in the last 12 months ) OR hormone-naive patients treated by surgery or external radiotherapy or brachytherapy for prostate adenocarcinoma but with persistent biological disease (PSA detectable after prostatectomy, or unchanged or increasing PSA after external radiotherapy or brachytherapy);
* Diagnostic recurrence assessment by any information or examination carried out since the ascension of the PSA, not having revealed local recurrence or lymph node lesions which may benefit from to external radiation
* Signed informed consent.

Exclusion Criteria:

* Patient already treated by hormonotherapy;
* Formal contraindication to hormonotherapy;
* Formal contraindication to external radiotherapy
* Formal contraindication to the Lasilix administration during the PET exams: Hypersensitivity to Furosemide or to one of the excipients, functional acute renal insufficiency, hepatic encephalopathy, urinary tracts obstruction, hypovolemia or dehydration, severe hypokalemia, severe hyponatremia, hepatitis in evolution and severe hepatocellular insufficiency in haemodialysis patient and patient presenting a severe renal insufficiency (creatinine clearance <30 ml / min) due to the risk of accumulation of furosemide, which is then mainly eliminated by the biliary route;
* Significant cardiovascular affection such as myocardial infarction within the last 6 months preceding inclusion, severe rhythm disturbances, stroke within 6 months prior to inclusion, prolonged corrected QT interval with QTc > 450 msecs according to Bazett formula;
* Impossibility to comply with the study follow-up for geographical or psychic reasons.
* Patient under protection of justice (Under tutorship, curatorship or deprived of liberty)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of patients presenting a positive PET during the initial PSMA-PET (prior to androgenic blockade) and the PSMA-H-PET (PSMA PET after androgenic blockade), patient being his own witness | Day 14 after the androgenic blockade
  PSMA-PET

SECONDARY OUTCOMES:
Evaluation of the reproductibility of the PSMA-PET and PSMA-H-PET interpretation | Day 14 after the androgenic blockade
  PSMA-PET and PSMA-H-PET
Evaluation of the impact of androgenic blockade on lesions revealed by PSMA-H PET in comparison with the initial PSMA-PET | Day 14 after the androgenic blockade
  Number of lesions (PSMA-ET and PSMA-H PET)
Evaluation of the impact of androgenic blockade on lesions revealed by PSMA-H PET in comparison with the initial PSMA-PET | Day 14 after the androgenic blockade
  Fixation intensity (PSMA-ET and PSMA-H PET)
Evaluation of the PSMA-PET and PSMA-H PET impact in the therapeutic management modifications | Day 14 after the androgenic blockade
  Comparison between treatments planned after PSMA-PET and treatments planned after PSMA-H-PET
Evaluation of the interest of late pelvic acquisition 3 hours after the PSMA-68Ga injection | Day 14 after the androgenic blockade
  PSMA-PET and PSMA-H-PET efficience
Evaluation of the results correlation of each PSMA-PET with clinical data, histologic primary tumor and biologic data of the recurrence (PSA kinetic and velocity assessed at screening) | Day 14 after the androgenic blockade
  PSMA-PET efficience
Evaluation of the results correlation of each PSMA-PET with clinical data, histologic primary tumor and biologic data of the recurrence (PSA kinetic and velocity assessed at screening) | Day 14 after the androgenic blockade
  PSA rate
Evaluation of the correlation between the PSA and testosterone rates variations between D0 and D14 and the PSMA-PET results | Day 14 after the androgenic blockade
  PSA and testosterone rates and PSMA-PET results
Tolerance profile | Up to Day 15-30 visit
  Incidence of PSMA-H-PET Adverse Events assessed by the Common Terminology Criteria for Adverse Events (CTCAE version 5.0)

OTHER OUTCOMES:
In case of envisaged irradiation, impact on the modifications of irradiation volumes between the initial PET-PSMA and the PET-PSMA-H | Day 14 after the androgenic blockade
  PET-PSMA and PET-PSMA-H

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure GIRAUDET, MD, Principal Investigator — Centre Leon Berard; David KRYZA, MD, Principal Investigator — Centre Leon Berard
Locations (6):
- France (6):
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier de Grenoble Hôpital Nord Michallon, La Tronche
  - Centre Léon Bérard, Lyon
  - APHM - Hôpital Nord, Marseille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite